CLINICAL TRIAL: NCT00636064
Title: A Double-Blind Multicenter Study of the Safety and Efficacy of Parecoxib Sodium/Valdecoxib and Placebo/Valdecoxib Compared to Placebo for Treatment of Post-Surgical Pain in Patients Who Have Coronary Bypass Graft Via Median Sternotomy
Brief Title: A Study Comparing the Efficacy and Safety of Valdecoxib Plus Parecoxib Versus Valdecoxib Plus Placebo for the Treatment of Pain After Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PARA-0505-071; A3481015
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — parecoxib; valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: Parecoxib Sodium/Valdecoxib
- B (Experimental)
  Interventions: Drug: Placebo/Valdecoxib
- C (Experimental)
  Interventions: Other: Placebo/Placebo

INTERVENTIONS:
Drug: Parecoxib Sodium/Valdecoxib — Parecoxib sodium 40 mg intravenous (IV) on the day after surgery (Day 1) following recovery from anesthesia, contingent on an acceptable postoperative status, verification of baseline eligibility, and lack of perioperative complications. A second dose of parecoxib sodium 20 mg IV was administered on Day 1. On the day following surgery, patients received parecoxib 20 mg IV at 8 am and each subsequent dose was administered at 12-hour intervals. After receiving at least 6 doses of IV parecoxib sodium, patients were transitioned to oral valdecoxib 20 mg taken at 12-hour intervals until the total treatment duration of 10 days had been completed.
  Arms: A
Drug: Placebo/Valdecoxib — Patients received placebo matched to parecoxib sodium 40 mg IV on Day 1 following recovery from anesthesia, contingent on an acceptable postoperative status, verification of baseline eligibility, and lack of perioperative complications. A second dose of placebo matched to parecoxib sodium 20 mg IV was administered on Day 1. On the day following surgery, patients received placebo matched to parecoxib sodium 20 mg IV at 8 am and each subsequent dose was administered at 12-hour intervals. After receiving at least 6 doses of IV placebo, patients were transitioned to oral valdecoxib 20 mg taken at 12-hour intervals until the total treatment duration of 10 days had been completed.
  Arms: B
Other: Placebo/Placebo — Patients received placebo matched to parecoxib sodium 40 mg IV on Day 1 following recovery from anesthesia, contingent on an acceptable postoperative status, verification of baseline eligibility, and lack of perioperative complications. A second dose of placebo matched to parecoxib sodium 20 mg IV was administered on Day 1. On the day following surgery, patients received placebo matched to parecoxib sodium 20 mg IV at 8 am and each subsequent dose was administered at 12-hour intervals. After receiving at least 6 doses of IV placebo, patients were transitioned to oral placebo matched to valdecoxib 20 mg taken at 12-hour intervals until the total treatment duration of 10 days had been completed.
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of parecoxib/valdecoxib therapy and placebo/valdecoxib therapy for the treatment of pain after coronary artery bypass surgery

ELIGIBILITY:
Inclusion criteria:

* Patients expected to receive in-hospital pain medication for pain after coronary artery bypass graft surgery for at least 3 full days and pain medication over a 10-day period
* New York Heart Association Class I to III or cardiac ejection fraction of at least 35% before surgery
* Body mass index of less than or equal to 40 kg/m2 and weight of >55 kg
* Patients scheduled to undergo an isolated (bypass grafting only without valve replacement, significant aortic reconstruction, or ventriculoplasty) primary CABG surgery via median sternotomy, using cardiopulmonary bypass

Exclusion criteria:

* Patient has undergone or is going to have emergency coronary artery bypass graft surgery or surgery without cardiopulmonary bypass procedure
* Symptomatic peripheral vascular disease
* Heart attack within 48 hours of surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1671 (Actual)
Dates: Start 2003-01; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Combined incidence of the number of patients with at least 1 confirmed clinically relevant adverse event (CRAE) | Day 30

SECONDARY OUTCOMES:
Combined incidence of the number of patients with at least 1 reported CRAE and the combined incidence of the number of patients with specific reported CRAEs summarized according to the categories listed above | Day 30
Rate of supplemental analgesia consumed | Days 1-10
Vital signs | Day 30
Summed Pain Intensity (SPI) of sternotomy alone and overall body pain over 8 hours (SPI 8) | Day 1
Opioid-related Symptoms Distress Scale (OR-SDS) | Days 1-10
Time to last Patient Controlled Analgesia (PCA) dose
Recovery measures (length of stay, intensive care unit/hospital recovery and eligibility for discharge)
Combined incidence of the number of patients with specific confirmed CRAEs in categories of cardiovascular thromboembolic CRAEs, renal CRAEs, upper gastrointestinal ulcer CRAEs, and wound healing complication CRAEs | Day 30
Adverse events | Day 30
Serious adverse events | Day 30
Clinical laboratory assessments | Day 30
Peak Pain Intensity (PPI) of sternotomy alone and overall body pain | Days 1-10
Patient's and Physician's Global Evaluation of Study Medication | At time of transition from intravenous to oral medication and final visit/early termination
Modified Brief Pain Inventory-short form (mBPI-sf) | Days 1-10
SPI of sternotomy alone and overall body pain over 12 hours (SPI 12) and 24 hours (SPI 24) | Days 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (160):
- United States (64):
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Springdale, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Fort Collins, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Hudson, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Salisbury, Maryland
  - Pfizer Investigational Site, Takoma Park, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Cambridge, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Muskegon, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Sandusky, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Amarillo, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Falls Church, Virginia
  - Pfizer Investigational Site, Fredericksburg, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Elkhorn, Wisconsin
  - Pfizer Investigational Site, Madison, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - Pfizer Investigational Site, Morón, Pcia. de Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Australia (3):
  - Pfizer Investigational Site, Auchenflower, Queensland
  - Pfizer Investigational Site, Ashford, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
- Pfizer Investigational Site, Graz, Austria
- Belgium (4):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Liège
- Canada (11):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Fleurimont, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Colombia (4):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Floridablanca, Santander Department
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
  - Pfizer Investigational Site, Bogotá
- Czechia (2):
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Prague
- Denmark (2):
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Odense C
- Finland (3):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Turku
- Germany (10):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Giessen
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
- Pfizer Investigational Site, Dublin, Ireland
- Israel (9):
  - Pfizer Investigational Site, Beersheba
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Holon
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Ramat Gan
  - Pfizer Investigational Site, Rehovot
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (4):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pisa
- Mexico (3):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Mexico City, Mexico DF
  - Pfizer Investigational Site, Mexico City, Mexico, DF
- Netherlands (3):
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Zwolle
- Pfizer Investigational Site, Feiring, Norway
- Poland (5):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Romania (3):
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Cluj-Napoca
  - Pfizer Investigational Site, Timișoara
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Singapore, Singapore
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
- South Africa (8):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Les Marais, Pretoria
  - Pfizer Investigational Site, Parow, Western Cape
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Pretoria
- Spain (3):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- Switzerland (2):
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
- United Kingdom (5):
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Middlesbrough
  - Pfizer Investigational Site, Oxford

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PARA-0505-071&StudyName=A%20study%20comparing%20the%20efficacy%20and%20safety%20of%20valdecoxib%20plus%20parecoxib%20versus%20valdecoxib%20plus%20placebo%20for%20the%20treatment%20of%20pain%20a